CLINICAL TRIAL: NCT04098861
Title: Efficacy and Safety of Latanoprost/Timolol Fixed Combination Dosed Twice Daily Compared to Once Daily in Patients With Primary Open Angle Glaucoma
Brief Title: Efficacy and Safety of Latanoprost/Timolol for Primary Open Angle Glaucoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Norshamsiah Md Din, Associate Professor, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FF-2019-058
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost; Timolol

STUDY DESIGN:
Intervention Model Description: A single-center, randomized open-labeled, prospective, crossover study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- once daily group (Experimental): Latanoprost/Timolol Fixed Combination (LTFC) will be administered once daily for 4 weeks. The IOP will be determined on Day 14 and 28. The following examinations will be performed: evaluation of conjunctiva hyperemia, anterior chamber reaction, applanation tonometry, measurement of blood pressure and heart rate.
  For once daily dosing, the eye drops will be instilled at 8am every morning. The IOP will be taken at 9am-12pm on study day.
  Interventions: Drug: Latanoprost/Timolol
- twice daily group (Experimental): Latanoprost/Timolol Fixed Combination (LTFC) will be administered twice daily for 4 weeks. The IOP will be determined on Day 14 and 28. The following examinations will be performed: evaluation of conjunctiva hyperemia, anterior chamber reaction, applanation tonometry, measurement of blood pressure and heart rate.
  For twice dosing, the eye drops will be instilled at 8am and 8pm. The IOP will be taken at 9am-12pm on study day.
  Interventions: Drug: Latanoprost/Timolol

INTERVENTIONS:
Drug: Latanoprost/Timolol — Latanoprost/Timolol Fixed Combination

SUMMARY:
Intraocular pressure (IOP) is the most important modifiable risk factor to prevent and delay progression of glaucoma. IOP reduction has been proven to delay the onset and progression of glaucoma, and uncontrolled IOP is constantly associated with progression of visual field loss.

Medical therapy is the first line in IOP reduction for Primary Open Angle Glaucoma (POAG). It is a known fact that glaucoma patients often require addition of a second antiglaucoma medications when disease progresses or tachyphylaxis occurs. It was reported that more than 50% of patients require 2 or more medications to achieve optimum IOP control.

Nevertheless, compliance and adherence are often impaired with multiple-drug therapy. Combining two ocular hypotensive agents in one bottle may help patients adhere to therapeutic regimen by reducing the number of medications used and the total number of doses administered.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Able to provide informed consent
3. Diagnosed as having unilateral or bilateral, mild to moderate POAG
4. The POAG treated with only two antiglaucoma

Exclusion Criteria:

1. Advanced POAG
2. Patient with contraindication for topical use of a-blocker and prostaglandin analogue
3. Patient with contraindication for systemic use of a-blocker
4. Patient on systemic use of a-blocker such as metoprolol, propranolol, atenolol
5. History of orbital or ocular trauma.
6. History of cataract surgery less than 6 months.
7. History of previous ocular surgery; e.g. vitreoretinal surgery, corneal transplantation or glaucoma surgery
8. Any active eye infections or corneal ulceration.
9. Patient with ocular surface disease
10. Other ocular disease that might interfere with IOP measurements or result
11. Precious eye i.e patient with only one good eye
12. Contact lens is not allowed within 1 week before the start of study and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Enrollment: 40 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Intraocular pressure reduction | 4 weeks
  IOP reduction with LTFC given once and twice daily in POAG patients

SECONDARY OUTCOMES:
Safety: Side effects | 4 weeks
  Side effects of LTFC given twice daily in POAG patients

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided